CLINICAL TRIAL: NCT06464510
Title: Norepinephrine and Vasopressin for Rescue Versus Early Vasopressin for Vasopressor Dependent Sepsis: An Open-label, Multicenter, Randomized, Controlled Trial: NoVa
Brief Title: Norepinephrine and Vasopressin for Rescue Versus Early Vasopressin for Vasopressor Dependent Sepsis
Acronym: NoVa
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Brazilian Research in Intensive Care Network (BRICNet) (Unknown); National Institute of Science and Technology (INCT) in Precision Intensive Care Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ip_hcor_nova
Record Dates: First submitted 2024-06-11; First posted 2024-06-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-03

CONDITIONS: Septic Shock
Keywords: Vasopressin; Norepinephrine; Vasopressor dependent sepsis; Septic shock; Critically ill
MeSH Terms: conditions — Shock, Septic; Diabetes Insipidus; Critical Illness | interventions — Norepinephrine; Vasopressins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Vasopressin (Experimental): After randomization, vasopressin will be initiated and titrated up to 0.04U/min to maintain the target mean arterial pressure (MAP). Concurrently, norepinephrine will be reduced, with the goal of using the maximum dose of vasopressin and minimizing or eliminating the use of norepinephrine, while still maintaining the target MAP.
  Interventions: Drug: Early Vasopressin
- Norepinephrine plus vasopressin for rescue (Active Comparator): After randomization, norepinephrine will be titrated to maintain the target MAP. Vasopressin will be introduced as a rescue strategy only if the norepinephrine dose exceeds 0.5 μg/kg/min. Once vasopressin is initiated, it can be titrated up to 0.04U/min to help maintain the target MAP if the norepinephrine dose remains above 0.5 μg/kg/min.
  Interventions: Drug: Norepinephrine and Vasopressin for Rescue

INTERVENTIONS:
Drug: Early Vasopressin — Early Vasopressin group: Vasopressin up to 0.04U/min initiated after randomization.
  Arms: Early Vasopressin
Drug: Norepinephrine and Vasopressin for Rescue — Norepinephrine and Vasopressin for Rescue group: Vasopressin up to 0.04U/min initiated only if norepinephrine dose exceeds 0.5 μg/kg/min.
  Arms: Norepinephrine plus vasopressin for rescue

SUMMARY:
The norepinephrine and vasopressin for rescue versus early vasopressin for vasopressor dependent sepsis (NoVa) is a phase 3, multicenter, open-label, randomized controlled trial comparing an early vasopressin initiation strategy versus norepinephrine plus vasopressin initiation only as a rescue strategy for hemodynamic management of critically ill patients with vasopressor dependent sepsis.

DETAILED DESCRIPTION:
Sepsis is defined as a life-threatening organ dysfunction caused by a dysregulated body response to infection. Its most severe form, septic shock, occurs when underlying circulatory and cellular metabolic abnormalities are pronounced, indicating greater severity and higher mortality. Vasopressor use is a cornerstone aspect in the treatment of critically ill patients with sepsis-associated hemodynamic dysfunction, with norepinephrine, a catecholamine, being the vasopressor of choice.

Vasopressin is an endogenous peptide hormone with potential advantages over norepinephrine in a catecholamine-sparing strategy for treating sepsis-associated hemodynamic dysfunction.

This is a phase 3, multicenter, open-label, randomized controlled trial. Adult patients with sepsis-associated hemodynamic dysfunction in the ICU may be eligible to participate. We aim to enroll 2,800 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vasopressor dependent sepsis, defined by infection suspicion and antibiotic administration or laboratory confirmed viral infection, plus hypotension with the need of vasopressors for at least one hour;
* Admitted or expected to be admitted to the ICU in the next 12 hours
* Adequate volume resuscitation in the opinion of the attending physician
* Use of norepinephrine > 0.05μg/Kg/min and ≤ 0.25μg/Kg/min for at least 1 hour and at most 24 hours at the time of inclusion

Exclusion Criteria:

* Use of norepinephrine > 0.25μg/Kg/min in the last 24 hours, except when administered transiently in the context of sedation for a procedure or the initial phase of volume resuscitation for a period of less than one hour
* Dialysis-dependent chronic kidney disease or acute kidney injury that received renal replacement therapy during current hospitalization or are expected to receive renal replacement therapy in the next 24 hours
* Use of other vasopressors (except norepinephrine) at the moment of inclusion
* Use of vasopressors for sepsis in the last 7 days
* Suspected or confirmed acute mesenteric ischemia
* Anaphylaxis or known hypersensitivity to the study drug
* Expect to die in the next 24 hours
* Medical team not committed to full support at the time of inclusion
* Previous inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2800 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality or renal replacement therapy | 28 days
  Composite of all-cause mortality or renal replacement therapy within 28 days after randomization.

SECONDARY OUTCOMES:
All-cause mortality | 28 days
  All-cause mortality within 28 days after randomization
Renal replacement-therapy | 28 days
  Need of renal replacement therapy within 28 days after randomization.
Renal replacement-free days | 28 days
  Renal-replacement free days are defined by the number of days a patient is alive and free of renal replacement support between randomization and day 28. Non-survivors will be considered to have zero renal replacement-free days.
ICU-free days | 28 days
  Number of days a patient is alive and outside the ICU between randomization and day 28. Non-survivors will be considered to have zero ICU-free days.
Hospital-free days | 28 days
  Number of days a patient is alive and outside the hospital between randomization and day 28. Non-survivors will be considered to have zero hospital-free days.
Organ support-free days and its components | 28 days
  The definition of organ support involves three components: renal replacement therapy, invasive mechanical ventilation, and vasopressor use.
  Organ support-free days are defined by the number of days a patient is alive and free of all three organ support therapies between randomization and day 28. Non-survivors will be considered to have zero organ support-free days.
Cardiac arrhythmias | 28 days
  Occurrence of cardiac arrhythmias between randomization and day 28
Ischemic events | 28 days
  Occurrence of mesenteric ischemia, ischemic stroke, digital ischemia and acute coronary syndrome between randomization and day 28

CONTACTS AND LOCATIONS:
Overall Officials: Bruno M Tomazini, MD, Principal Investigator — Hcor Research Institute; Machado R Flavia, PhD, Study Chair — Universidade Federal de São Paulo
Locations (8):
- Brazil (8):
  - Hospital Geral de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Hospital Nereu Ramos, Florianópolis, Santa Catarina
  - Hospital SEPACO, São Paulo, S
  - Hospital de Amor - Unidade Barretos (Fundação PIO XII), Barretos, São Paulo
  - Hospital do Coracao, São Paulo, São Paulo
  - BP-A Beneficiência Portuguesa de São Paulo, São Paulo, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Hospital São Paulo - UNIFESP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Submission of a statistical analysis plan for the purposed analyses for the Steering Committee evaluation. Compliance with Brazilian data privacy law.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after study publication
Access Criteria: Submission of a statistical analysis plan for the purposed analyses for the Steering Committee evaluation. Compliance with Brazilian data privacy law.